CLINICAL TRIAL: NCT06283953
Title: Boosting Resources and Caregiver Empowerment for Trach Care at Home: A Pragmatic Randomized Trial
Brief Title: Boosting Resources for Tracheostomy Care at Home
Acronym: BREATHE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital of Philadelphia (Other); Children's Hospitals and Clinics of Minnesota (Other); Children's National Research Institute (Other); Rady Children's Hospital, San Diego (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023P001695; IHS-2022C1-26100 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Tracheostomy; Caregiver Burden
Keywords: shared decision making; patient reported outcomes; tracheostomy; ventilator; caregiver; discharge program; pediatric
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of care team delivering the interventions and of caregiver participants receiving the interventions is not possible for this study.
  The outcome assessors collecting the readmission data and statistician conducting analyses will be blinded to the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active Comparator Caregivers (Active Comparator): TrachMeHome program delivered in the hospital including education, skills training and case management for caregivers
  Interventions: Behavioral: Trach Me Home
- Intervention Caregivers (Experimental): Trach Me Home and Trach Plus with additional education, outpatient care team communication and social support for caregivers.
  Interventions: Behavioral: Trach Plus; Behavioral: Trach Me Home
- Active Comparator Physicians (Active Comparator): Primary care physicians' of the enrolled participant's child receiving discharge communication
  Interventions: Behavioral: Trach Me Home
- Intervention Physicians (Experimental): Primary care physicians' of the enrolled participant's child receiving outpatient care team communication prior to discharge
  Interventions: Behavioral: Trach Plus; Behavioral: Trach Me Home

INTERVENTIONS:
Behavioral: Trach Plus — The Trach Plus program includes education, social support, and outreach to outpatient care team.
  Arms: Intervention Caregivers; Intervention Physicians
Behavioral: Trach Me Home — The Trach Me Home discharge program includes caregiver education, skills training and case management.

SUMMARY:
The goal of this trial is to advance the understanding of how to best support caregivers of children with tracheostomies who are caring for their child at home. The main questions it aims to answer are:

* What are the best ways to support caregivers post-discharge with both medical and nonmedical decisions about resuming life, work, and family activities, while safely caring for their child with a tracheostomy at home?
* How can the investigators leverage existing technology to facilitate communication between inpatient and outpatient care teams to better support needs of pediatric patients and caregivers post-discharge?

Caregiver participants will be randomly assigned to receive Trach Me Home (gold standard discharge program) or Trach Me Home with additional components. Caregiver participants will complete three surveys over the course of 6 months. Researchers will see if caregivers in the Trach Me Home with additional components report lower caregiver burden at 4 weeks post discharge (primary outcome) and fewer hospital readmissions at 6 months than those in Trach Me Home arm.

DETAILED DESCRIPTION:
The study is focused on a rare and medically complex population of children with tracheostomies. The study is a Type I hybrid effectiveness-implementation study using a pragmatic randomized trial at six participating sites. The goal of this trial is to advance the understanding of how to best support caregivers of children with tracheostomies who are caring for their child at home. The main question[s] it aims to answer are:

* What are the best ways to support caregivers post-discharge with both medical and nonmedical decisions about resuming life, work, and family activities, while safely caring for their child with a tracheostomy at home?
* How can the investigators leverage existing technology to facilitate communication between inpatient and outpatient care teams to better support needs of pediatric patients and caregivers post-discharge?

Caregiver participants will randomly assigned to the Comparator arm (gold standard discharge program) or to the Intervention arm (gold standard program with other components). Caregiver participants will complete three surveys over the course of 6 months. The investigators will test two main hypotheses: the Intervention arm will have (1) significantly lower caregiver burden at 4 weeks post discharge (primary outcome) and (2) significantly lower readmissions or emergency room visits at 6 months post discharge than the Comparator arm.

The investigators will also survey pediatricians of participating patients at 6 months post discharge and examine whether intervention arm pediatricians have higher satisfaction with discharge communication than those in comparator arm.

ELIGIBILITY:
Inclusion Criteria:

* Lead or primary adult caregiver (18 or older) of infants or children (0-17 years old) with tracheostomy who are planning for discharge to home, including children who are dependent on ventilator

Exclusion Criteria:

* Patients transferred to other hospital or facility (and/or not discharged to home during study period)
* Primary caregiver unable to read or write in English, Spanish, Mandarin, or Arabic
* Not residing in the U.S. for at least 12 months after discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden | 4 weeks post-discharge
  Pediatric Tracheostomy Health Status Instrument (PTHSI) Caregiver burden subscale, total scores range from 0-68. Higher scores indicate higher burden.

SECONDARY OUTCOMES:
Medical Complications Associated with Tracheostomy | 6 months post-discharge
  4-item modified Medical Complications Associated with Tracheostomy (MCAT) measure that includes 4 caregiver reported items to assess the total number of urgent medical visits, emergency room and readmissions for tracheostomy-related issues. Items are summed and scores start at 0 and there is no upper limit. Higher total numbers are worse.
6-month Readmission Rate | 6 months post-discharge
  Percentage with one or more emergency room visits or hospital readmissions as documented in the electronic health record within 6 months of discharge.
Frequency of pediatrician communication | 6 months post-discharge
  Percentage of pediatrician-specific communication with inpatient team prior to and/or shortly after discharge documented in electronic medical record or by pediatrician report.
Primary care pediatrician satisfaction | 6 months post-discharge
  Clinician reported satisfaction with discharge communication scored from 0-100, higher scores indicate higher satisfaction with discharge communication.
Medical Complications Associated with Tracheostomy | 4 weeks post-discharge
  4-item modified Medical Complications Associated with Tracheostomy (MCAT) measure that includes 4 caregiver reported items to assess the total number of urgent medical visits, emergency room and readmissions for tracheostomy-related issues. Items are summed and scores start at 0 and there is no upper limit. Higher total numbers are worse.
Caregiver Burden | 6 months post-discharge
  Pediatric Tracheostomy Health Status Instrument (PTHSI) Caregiver burden subscale, total scores range from 0-68. Higher scores indicate higher burden.

OTHER OUTCOMES:
Number of readmissions | 6 months post discharge
  The total number of electronic health record documented emergency room visits and hospital admissions will be collected, with higher numbers being worse (indicating more readmissions).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital; Christopher Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary / Massachusetts General Hospital
Locations (6):
- United States (6):
  - University of San Diego Rady Children's Hospital, La Jolla, California
  - Children's National Medical Center, Children's Research Institute, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
To promote research replicability, transparency and future use of the data, de-identified data sets will be created and will be available, by request, to outside researchers.
  The Data Package (comprised of the de-identified Analyzable Data Set, Full Protocol, metadata, data dictionary, full statistical analysis plan, and analytic code from the project) will be deposited in the Patient-Centered Outcomes Research Institute's Data Repository at the ICPSR. Participant information sheets for the study will indicate that de-identified information will be deposited in an open access service to promote use of the data by other researchers. No information that contains identifiers or that could be used to link an individual to the data will be included in the de-identified data set. No data will be provided from qualitative transcripts as this may lead to identifying information about participants. However, codes abstracted from qualitative transcripts may be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study results have been published, about 1 year after the end of the funded grant period, the study materials and de-identified data will be placed on an open access service such as ICPSR where they will be available indefinitely.
Access Criteria: Researchers may access the data through the PCORI-designated repository (ICPSR's website) once it is made available.

REFERENCES:
- [Derived] Sepucha K, Callans K, Leavitt L, Chang Y, Vo H, Brigger M, Broughton S, Cahill J, Chinnadurai S, Germann J, Giordano T, Greenlick-Michals H, Javia L, Jayawardena ADL, Osthimer J, Patel RC, Redmann A, Roumiantsev S, Simmons L, Smith M, Tate M, Warren M, Whalen K, Yager P, Zalzal H, Hartnick C. Boosting REsources And caregiver empowerment for Tracheostomy care at HomE (BREATHE) Study: study protocol for a stratified randomization trial. Trials. 2024 Oct 28;25(1):722. doi: 10.1186/s13063-024-08522-x. PMID 39468582